CLINICAL TRIAL: NCT04403841
Title: Effect of Group Patient Education on Glycemic Control Among People Living With Type 2 Diabetes in Vietnam: a Randomized Controlled Trial
Brief Title: Effect of Group Patient Education on Glycemic Control Among People Living With Type 2 Diabetes in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Ho Thi Kim Thanh, Associate Professor, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HMU16227
Record Dates: First submitted 2020-05-14; First posted 2020-05-27 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; education; glycemic
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The intervention of group education on type 2 diabetes, including, in addition to usual diabetes care
  Interventions: Other: patient education and self-management intervention in a low-resource setting on diabetes knowledge and levels of blood glucose control
- Control (Other): Patients meeting the inclusion criteria assigned to usual diabetes care alone
  Interventions: Other: Usual diabetes care alone

INTERVENTIONS:
Other: patient education and self-management intervention in a low-resource setting on diabetes knowledge and levels of blood glucose control — The intervention consisted group education on type 2 diabetes, including, in addition to usual diabetes care: information on diet, exercise, drug therapy, and adherence
  Arms: Intervention
Other: Usual diabetes care alone — Usual diabetes care was consistent with the ADA guidelines (15) and comprised standard dietary and exercise advice in addition to antidiabetes treatment
  Arms: Control

SUMMARY:
This study measures the effect of a 3-month patient education and self-management intervention in a low-resource setting, on diabetes knowledge and levels of blood glucose control.

DETAILED DESCRIPTION:
In Vietnam, there is a low level of diabetes knowledge among the general population, and significantly lower awareness in rural areas compared with urban areas. This highlights the urgent need for communication and education to improve the knowledge of the Vietnamese population of patients with type 2 diabetes on risk factors, complications, prevention and treatment. The main goal of this study is to evaluate the effects of a patient education and self-management intervention as add-on to usual diabetes care in a low-resource setting on diabetes knowledge and blood glucose control parameters in Vietnamese patients with type 2 diabetes.

This is a single-center, randomized, controlled study among adult out-patients with type 2 diabetes. Patients meeting the inclusion criteria are randomly assigned to a community intervention or to usual diabetes care alone (control group) for a period of 3 months. The intervention consists of group education on type 2 diabetes, including, in addition to usual diabetes care: information on diet, exercise, drug therapy, and adherence. Each patient should attend the group education monthly over 3 consecutive months. Usual diabetes care is consistent with the ADA guidelines and comprises standard dietary and exercise advice in addition to antidiabetes treatment. Diabetes knowledge is measured with a modified Michigan University Diabetes Knowledge Test (MDKT). Other study outcomes includes change in mean HbA1c, fasting blood glucose, and systolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes as defined above
* Aged 40-80 years old
* Ability to attend monthly clinic visits and signed informed consent
* All antidiabetes treatments were permitted including insulin

Exclusion Criteria:

* A diagnosis of mental or neurological diseases that could interfere with the ability to comply with study procedures
* Pregnancy or lactation
* Known drug or alcohol dependence
* Requirement for a change in antidiabetes treatment over the study period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Disease awareness | 3-month
  All patients complete a modified Michigan University Diabetes Knowledge Test (MDKT) (16) at baseline and at the end of the 3-month trial. The MDKT is a quick and low-cost method of assessing general knowledge of diabetes and diabetes self-care. The 23-item original questionnaire was translated into Vietnamese and adapted as required based on a pilot test performed in 10 people with type 2 diabetes, which resulted in one question being removed. The modified questionnaire therefore consist of 22 statements with multiple choice answers with 1 point awarded for each correct answer (Appendix 1). Patients who answer >50% of the questions correctly considered to pass the knowledge test, and patients who answer <50% of the questions correctly considered to fail. The proportion of successful patients (i.e. with MDKT total score ≥11) the study primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thanh HTK, Tien TM. Effect of Group Patient Education on Glycemic Control Among People Living with Type 2 Diabetes in Vietnam: A Randomized Controlled Single-Center Trial. Diabetes Ther. 2021 May;12(5):1503-1521. doi: 10.1007/s13300-021-01052-8. Epub 2021 Apr 11. PMID 33840068